CLINICAL TRIAL: NCT02865018
Title: An Open Label, add-on Trial of Cetirizine for Patients With Neuromyelitis Optica
Brief Title: Neuromyelitis Optica (NMO) & Cetirizine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Guthy Jackson Charitable Foundation (Other)
Responsible Party: Principal Investigator, Ilana Katz Sand, Assistant Professor of Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1513
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Neuromyelitis Optica
Keywords: Neuromyelitis Optica; Cetirizine
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetirizine (Experimental): 10mg oral each day
  Interventions: Drug: cetirizine

INTERVENTIONS:
Drug: cetirizine
  Other Names: Zyrtec

SUMMARY:
Neuromyelitis optica (NMO) is an autoimmune disease that affects the central nervous system. Patients have relapses (also known as attacks) which are often quite severe and leave them with significant disability. Without treatment, within 5 years 50% of NMO patients are blind in one or both eyes or require walking assistance (cane, walker or wheelchair).

NMO has only been relatively recently described and is fairly rare. Most NMO patients' immune systems produce abnormal antibodies against aquaporin-4 (AQP4), which is found in certain cells in the central nervous system. When these AQP4 antibodies bind to AQP4, they trigger a cascade of events involving the immune system which eventually leads to damage to the nervous system. This ultimately leads to disability, some of which is permanent.

Until now, treatments for NMO have been mostly focused on decreasing production of this AQP4 antibody. However, recent experiments in animal models of NMO have shown the importance of what happens inside the central nervous system after the antibody binds to the nervous system cell. Specifically, researchers have noted the importance of a specific cell type, eosinophils, in causing damage in NMO lesions. In a recent study, researchers showed they could prevent damage from NMO by blocking eosinophils using cetirizine, which is a popular over-the-counter allergy medicine.

Cetirizine is already known to be safe and well-tolerated in the general population. In this study, the researchers plan to add cetirizine on to patients' current NMO treatment. The researchers aim to show that it is safe, well-tolerated, and that with cetirizine, NMO patients have less relapses and therefore less disability over the course of the year following initiation of treatment. The researchers also plan to study how cetirizine changes the immunological profile in NMO patients by examining blood and cerebrospinal fluid.

DETAILED DESCRIPTION:
The researchers hypothesize that cetirizine, an allergy medication that acts as an eosinophil-stabilizer, will decrease the relapse rate when added to current standard therapy in patients with neuromyelitis optica.

Medication compliance will be assessed by the research coordinator at each visit through discussion with the patient and pill counting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 85
* Meet criteria for the diagnosis of neuromyelitis optica as outlined by Wingerchuk et al in 2006. Alternatively patients may be included if they have had an episode of myelitis or optic neuritis in combination with a positive NMO IgG antibody, as positive antibody with a first episode is highly associated with future relapse.
* Disease duration of at least 6 months
* Stable, without any NMO relapses, for the 3 months prior to the baseline assessment visit
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.

Exclusion Criteria:

* Current therapy with daily cetirizine or another daily antihistamine for any indication
* Known hypersensitivity to cetirizine, hydroxyzine, or any component of the formulation
* Change in NMO disease-modifying therapy in the 3 months prior to baseline assessment
* Pregnancy or planning pregnancy during the study period
* Severe renal or hepatic impairment
* Inability to complete the study protocol for any reason

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Katz Sand, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four potential participants were referred by treating physicians at the Corinne Goldsmith Dickinson Center for Multiple Sclerosis at Mount Sinai between April 2014 and February 2015. Sixteen were enrolled between Aprill 2014 and February 2016.
Groups:
- Cetirizine: 10mg oral each day for 1 year
Period: Overall Study
Arm/Group | Cetirizine
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cetirizine
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36.5 [27.1 to 51.0]
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age at Symptom onset | 31.0 [22.5 to 41.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 1
Positive NMO antibody in serum [Count of Participants; unit: Participants] | 13
Type of NMO Preventative Treatment at Enrollment [Count of Participants; unit: Participants]
  Rituximab | 8
  Azathioprine | 1
  Mycophenolate | 7
Duration of Current Treatment [Median (Inter-Quartile Range); unit: months] | 18.3 [7.8 to 40.1]
Number of Previous Preventative NMO treatment types [Count of Participants; unit: Participants]
  0 | 10
  1 | 5
  2 | 1
Oral Prednisone use at Enrollment [Count of Participants; unit: Participants] | 1
Total pre-study relapses [Median (Inter-Quartile Range); unit: relapses] — Relapses were defined as "patient-reported symptoms or objectively observed signs typical of an acute inflammatory demyelinating event in the CNS, with duration of at least 24 hours, in the absence of fever or infection."
  relapses | 3.0 [1.5 to 5.0]
Total pre-study relapses while on current preventative treatment [Median (Inter-Quartile Range); unit: relapses] | 0.0 [0.0 to 1.0]
Annualized Relapse Rate [Median (Inter-Quartile Range); unit: relapses per treatment year] — The pre-study annualized relapse rate (ARR) was calculated by taking the number of relapses each participant had experienced after the start of their current reported NMO preventative treatment, divided by the length of time (in years) they had been receiving this treatment.
  relapses per treatment year | 0.0 [0.0 to 0.7]

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate Before Cetirizine
Description: Relapses defined as "patient-reported symptoms or objectively observed signs typical of an acute inflammatory demyelinating event in the CNS, with duration of at least 24 hours, in the absence of fever or infection." The on study ARR was calculated as the number of relapses during the study divided by the length of time in the study.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: relapses per year
Arm/Group | Cetirizine
Number analyzed (Participants) | 15
relapses per year
  Baseline | 0.4 (0.80)
  1 year | 0.1 (0.24)

2. Secondary Outcome: Epworth Sleepiness Scale
Description: Sedation as measured by Epworth Sleepiness Scale. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score 0 to 24 from unlikelihood of abnormally sleep to excessively sleepy.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetirizine
Number analyzed (Participants) | 15
units on a scale
  Baseline | 6.5 (5.33)
  1 year | 6.9 (4.50)

3. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: Disability as measured by Expanded Disability Status Scale (EDSS). The EDSS provides a total score on a scale from 0 to 10, from normal function to lessening function with higher score, 10, being death due to MS.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetirizine
Number analyzed (Participants) | 15
units on a scale
  Baseline | 3.9 (2.18)
  1 year | 3.2 (2.31)

4. Secondary Outcome: Eotaxin Plasma Levels
Description: Eotaxin - an eosinophil-specific chemoattractant in the blood. Immunological measures related to eosinophil activity. Eotaxin plasma levels.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Cetirizine
Number analyzed (Participants) | 15
pg/mL | 19.25 [1.44 to 27.75]

ADVERSE EVENTS:
Arm/Group | Cetirizine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetirizine (N=15)
Unilateral eye pain with movement (Eye disorders) | 1
Blurry vision with difficulty distinguishing colors (Eye disorders) | 1
Neuro episode (Nervous system disorders) | 2 — re-emergence of old symptoms

LIMITATIONS AND CAVEATS:
Small sample size and lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes